CLINICAL TRIAL: NCT01901939
Title: Role of Exercise in Reversal of Hospitalization-associated Disability in Elderly
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Roberta Oka, Associate Chief Nurse for Research and Advanced Practice Nursing, Palo Alto Veterans Institute for Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OKR0003ADM
Record Dates: First submitted 2013-06-21; First posted 2013-07-17 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Aging
Keywords: exercise; elderly; activities of daily living; disability
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: observational
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Experimental): daily bedside tailored low intensity pedaling exercise
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — daily tailored low level pedaling exercise at bedside

SUMMARY:
The proposed preliminary study from this interdisciplinary team will provide important information about the feasibility and safety of bedside low intensity pedaling exercise during hospitalization. The findings from this study are essential to develop high-value, effective treatments that can be used by any hospital setting throughout the country. The program that investigators are proposing may provide important changes in how disability can be prevented in elderly patients who are hospitalized because of an acute illness.

DETAILED DESCRIPTION:
The study design includes 2 phases (10 months each) for development and evaluation of the testing and intervention protocol. The last 4 months of the study will be devoted to preparation of a larger randomized controlled clinical trial grant submission. Mixed methods will be used in both phases.

Phase I will focus on developing, testing and refining the measurement protocol and bedside tailored low intensity pedaling exercise (Ex) program using mixed methods. During this 10-month phase, researchers plan to enroll 10 participants who are admitted to a medical surgical (MS) unit and meet study eligibility criteria. Investigators will implement our proposed testing and intervention protocol,obtain feedback and make modifications as necessary. For this purpose the study team will use a process improvement framework with rapid cycle improvements. The outcome for Phase I will be development of a manual of operations for the testing and Ex protocol that will be implemented in Phase II.

Phase II (10 months) will randomly assign 60 patients over the age of 65 years who meet medical criteria and are admitted to a medical surgical (MS) hospital unit at the VA Palo Alto Health care system (VAPA HCS) to one of two groups, 1) low intensity bedside pedaling exercise or 2) usual care. All participants will be asked to complete questionnaires, undergo a Short Physical Performance Battery (SPPB), cognitive testing and a blood draw prior to participation in the Ex program (baseline). All testing and blood draw will be repeated within 24 hours prior to discharge (release from the hospital to home or other facility, indicating that their condition has been resolved or adequately treated or is stabilized during their hospital stay) from the hospital(approximately at 5-6 days). Participants will be followed for the duration of the hospital stay, an expected average length of 5-6 days. Additionally, all participants will be asked to continue to exercise after discharge to home for 4 weeks. All tests will be performed at baseline (prior to intervention), within 24 hours prior to discharge (release from the hospital to home or other facility, indicating that their condition has been resolved or adequately treated or is stabilized during their hospital stay)from the hospital, on average 5-6 days) and again at 4 weeks post discharge. The focus of Phase II is safety and feasibility of the intervention and association with outcome measures. The length of stay (LOS) at VAPA HCS is approximately 6 days. Thus, the study investigators anticipate that each individual will be enrolled approximately 5 days and participate in an average of 8 training sessions. Investigators will also examine the association between physical activity levels at baseline (pre Ex) and myokines and associated changes in myokines after intervention.

A description of the Ex program:

Individually tailored, low intensity bedside pedaling exercise:

Once participants complete the testing protocol they will be instructed in the bedside Ex program. Exercise intensity and duration will be individualized to the subject's physical limitations and tolerance. The PI is an Adult Nurse Practitioner (ANP), and will supervise and monitor exercise response including Heart Rate (HR), Blood Pressure (BP), Rating of Perceived Exertion (RPE), and symptoms (intensity, duration). Exercise will be terminated according to the American College of Sports Medicine (ACSM) criteria. Ex will consist of progressively increased pedaling exercise performed initially for one-two minutes, three times or more daily as tolerated. Pedaling exercise will be progressively increased as tolerated and appropriate. Cycle ergometry has been shown to be an effective exercise modality to maintain muscle strength and aerobic capacity in a variety of age groups. While inpatient exercise prescriptions utilize walking as the primary mode of exercise, recent studies show that despite known benefits of ambulation, multiple barriers prevent routine implementation in practice settings. The study investigators propose to examine the feasibility of a portable bedside pedaling device for exercise. This modality eliminates dependence on hospital staff to supervise ambulation and allows patients greater access to optimal treatment recommendations to maintain functional independence. This exercise modality is not new, but bedside use is novel. The pedaling device is sturdy and portable and will be placed at the foot of an anchored chair. Subjects will be able to pedal without fear of falling or interference from other devices. This exercise will be performed in addition to their normal ambulation requirements. All catheters and other devices will be secured so that accidental removal will not occur during the Ex session.

Adherence is a key component of this study and will be monitored during both phases of the pilot study. Adherence will be assessed by direct observation from PI/staff. Investigators will also examine potential barriers and facilitators to exercise training adherence by obtaining qualitative feedback from study participants. The qualitative information will provide greater depth of understanding to improve the delivery of the intervention as well as assist in optimizing adherence.

The Study team will also ask participants if they are willing to be contacted regarding future research that may be of interest to them.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* age 65 years or older
* Able to tolerate exercise
* Non-elective admission to hospital

Exclusion Criteria:

* Elective admission with expected LOS of 2 days or less
* Diagnosed with Dementia or Alzheimer's disease
* Lower extremity amputation
* Delirium
* Severe arthritis limiting ability to perform pedaling exercise
* Uncontrolled hypertension
* Hypotension
* Non-English speaking
* Participating in another clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Activities of Daily Living | Change from Baseline (Admission) to Discharge (approximately 3-5 days in length)
  Discharge is considered release from the hospital to home or other facility, indicating that their condition has been resolved or adequately treated or is stabilized during their hospital stay. On average we anticipate the time frame between hospital admission and discharge to be variable but between 3-5 days in length.

SECONDARY OUTCOMES:
Instrumental Activities of Daily Living | Change from Baseline (Admission) to Discharge (approximately 3-5 days in length)
  Discharge is release from the hospital to home or other facility, indicating that their condition has been resolved or adequately treated or is stabilized during their hospital stay. On average we anticipate the time frame between hospital admission and discharge to be variable but between 3-5 days in length.
Short Physical Performance Battery | Change from Baseline (Admission) to Discharge (approximately 3-5 days in length)
  Discharge is release from the hospital to home or other facility, indicating that their condition has been resolved or adequately treated or is stabilized during their hospital stay. On average we anticipate the time frame between hospital admission and discharge to be variable but between 3-5 days in length.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta K Oka, PhD, RN, Principal Investigator — VA Palo Alto HCS
Locations (1):
- VA Palo Alto HCS, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No